CLINICAL TRIAL: NCT03118765
Title: A Dose Ranging, Parallel Group, Active (Spiriva® Respimat®) And Placebo Controlled Study To Assess Relative Bioavailability, Pharmacodynamics And Safety Of Three Doses Of Tiotropium Bromide Inhalation Solution In Subjects With Mild To Moderate Chronic Obstructive Pulmonary Disease
Brief Title: Pharmacodynamic and Pharmacokinetic Dose Ranging Study of Tiotropium Bromide Administered Via Inhalation Solution in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glenmark Specialty S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSP304-201
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Mild to Moderate Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Test Treatment T1: GSP304 Inhalation Solution (Experimental)
  Interventions: Drug: GSP304 (tiotropium bromide) Inhalation Solution
- Test Treatment T2: GSP304 Inhalation Solution (Experimental)
  Interventions: Drug: GSP304 (tiotropium bromide) Inhalation Solution
- Test Treatment T3: GSP304 Inhalation Solution (Experimental)
  Interventions: Drug: GSP304 (tiotropium bromide) Inhalation Solution
- Test Treatment T4: GSP304 Placebo Inhalation Solution (Placebo Comparator)
  Interventions: Drug: GSP304 Placebo Inhalation Solution
- Test Treatment T5: Spiriva® Respimat® inhalation spray (Active Comparator)
  Interventions: Drug: Spiriva® Respimat® inhalation spray

INTERVENTIONS:
Drug: GSP304 (tiotropium bromide) Inhalation Solution — Once daily (QD) oral inhalation using a nebulizer
  Arms: Test Treatment T1: GSP304 Inhalation Solution; Test Treatment T2: GSP304 Inhalation Solution; Test Treatment T3: GSP304 Inhalation Solution
Drug: GSP304 Placebo Inhalation Solution — Once daily (QD) oral inhalation using a nebulizer
  Arms: Test Treatment T4: GSP304 Placebo Inhalation Solution
Drug: Spiriva® Respimat® inhalation spray — Once daily (QD) oral inhalation
  Arms: Test Treatment T5: Spiriva® Respimat® inhalation spray

SUMMARY:
Pharmacodynamic and Pharmacokinetic Dose Ranging Study of Tiotropium Bromide Administered Via Inhalation Solution in Patients With Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥40 years and ≤85 years of age at the time of consent.
* Subject must have a primary diagnosis of mild or moderate COPD defined as post-bronchodilator FEV1/FVC ratio of <70% and FEV1 of ≥50% of predicted normal value as per the NHANES III predicted normal values at screening.
* Willing to stop all other COPD medications or other medications which will interfere with the study results for the entire duration of the study, except albuterol/salbutamol as needed.
* Current or ex-smoker with ≥10 pack-year smoking history.

Exclusion Criteria:

* Subjects with a chest x-ray/CT scan that suggests a diagnosis other than COPD (eg, pneumonia, other infection, atelectasis, or pneumothorax or other active/ongoing pulmonary conditions) and taken within 6 months prior to study start. If there is no chest x-ray or CT scan taken within 6 months prior to study start, or if recent results are unavailable for review, a chest x-ray must be performed.
* Use of oral/parenteral corticosteroids or antibiotics for COPD within 6 weeks or depot corticosteroids within 3 months prior to screening or subject has had a change in dose or type of any medications for COPD within 14 days before screening.
* Hospitalization for COPD exacerbation or pneumonia within 3 months prior to screening.
* Subjects with a history of asthma, with the exception of outgrown childhood asthma, defined as transient wheezers outgrown by 5 years of age.
* Subject has a known history of alpha 1 antitrypsin deficiency-related emphysema.
* Subject requires nocturnal oxygen or continuous supplemental oxygen therapy.
* Subject with history of a positive result for HBsAg or HCV antibody.
* Subject is known to be seropositive for human immunodeficiency virus.
* Female subject is pregnant or lactating.
* Subject has a history of allergic reaction to the anti-cholinergic or any components of the study medications.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Caracta, MD FCCP, Study Director — Glenmark Pharmaceuticals
Locations (25):
- United States (25):
  - Glenmark Investigational Site 23, Andalusia, Alabama
  - Glenmark Investigational Site 12, Phoenix, Arizona
  - Glenmark Investigational Site 14, Tempe, Arizona
  - Glenmark Investigational Site 17, Fullerton, California
  - Glenmark Investigational Site 19, Edgewater, Florida
  - Glenmark Investigational Site 24, Miami, Florida
  - Glenmark Investigational Site 16, Miami, Florida
  - Glenmark Investigational Site 10, Miami Lakes, Florida
  - Glenmark Investigational Site 6, Orlando, Florida
  - Glenmark Investigational Site 20, Ormond Beach, Florida
  - Glenmark Investigational Site 21, Vero Beach, Florida
  - Glenmark Investigational Site 13, Winter Park, Florida
  - Glenmark Investigational Site 18, Las Vegas, Nevada
  - Glenmark Investigational Site 9, Charlotte, North Carolina
  - Glenmark Investigational Site 5, Columbus, Ohio
  - Glenmark Investigational Site 22, Columbus, Ohio
  - Glenmark Investigational Site 8, Dublin, Ohio
  - Glenmark Investigational Site 11, Medford, Oregon
  - Glenmark Investigational Site 3, Easley, South Carolina
  - Glenmark Investigational Site 2, Greenville, South Carolina
  - Glenmark Investigational Site 4, Greenville, South Carolina
  - Glenmark Investigational Site 1, Rock Hill, South Carolina
  - Glenmark Investigational Site 15, Spartanburg, South Carolina
  - Glenmark Investigational Site 7, Spartanburg, South Carolina
  - Glenmark Investigational Site 25, Tomball, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 155 subjects were randomized to study treatments.
Groups:
- GSP304 10 μg; GSP304 20 μg; GSP304 40 μg; Placebo; SPIRIVA RESPIMAT 5 μg: Oral inhalation, once daily (morning) for 21 days
Period: Overall Study
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg
Started | 30 | 32 | 31 | 32 | 30
Completed | 26 | 30 | 26 | 29 | 28
Not Completed | 4 | 2 | 5 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 1
Not completed — Non compliance with Study Procedures | 0 | 0 | 0 | 1 | 0
Not completed — Violation of Inclusion/ExclusionCriteria | 0 | 1 | 1 | 0 | 0
Not completed — COPD Exacerbation | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg | Total
Number analyzed (Participants) | 30 | 32 | 31 | 32 | 30 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (7.12) | 61.6 (10.34) | 65.4 (10.02) | 65.0 (9.51) | 62.0 (9.42) | 63.4 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 14 | 17 | 20 | 75
  Male | 17 | 21 | 17 | 15 | 10 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 4 | 1 | 2 | 12
  Not Hispanic or Latino | 28 | 29 | 27 | 31 | 28 | 143
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 7 | 2 | 1 | 1 | 13
  White | 27 | 25 | 29 | 31 | 29 | 141
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.848 (2.8936) | 26.150 (4.0007) | 24.799 (3.7138) | 25.409 (3.5321) | 25.503 (3.1809) | 25.543 (3.4803)

OUTCOME MEASURES:

1. Primary Outcome: Relative Bioavailability of Tiotropium With GSP304 in Comparison to SPIRIVA RESPIMAT 5 μg Based on CmaxSS
Description: The PK endpoint in plasma to assess the relative bioavailability was peak concentrations of tiotropium during the dosing interval at steady-state (CmaxSS)
Time Frame: Plasma concentrations on day 21 according to the below schedule: Pre-dose (0 hour), and at 2, 4, 6, 10, 15, 30, and 45, 60, 75, and 90 minutes post-dose, as well as 2, 4, 6, 8, 12, 16, 20 and 24 hours post-dose.
Population: The PK analysis set consisted of all subjects who were randomized, received at least 1 dose of study treatment, and had at least 1 quantifiable PK sample and did not have an exclusionary major protocol deviation.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 26 | 30 | 26 | 26
pg/mL | 4.10 (1.152) | 8.00 (1.140) | 21.80 (1.152) | 14.00 (1.152)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; GSP 304 vs SPIRIVA RESPIMAT 5 μg comparison for relative bioavailability data based on CmaxSS was tested and the estimated treatment ratios for the treatment comparisons was presented; Test type: Other — ANOVA; LS mean ratio (%) = 29.4, 90% CI 2-sided [21.14 to 41.00] — Relative Bioavailability (%) based on CmaxSS for of GSP304 in comparison to SPIRIVA RESPIMAT
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; [analysis description as in outcome 1, analysis 1]; Test type: Other — ANOVA; LS mean ratio (%) = 57, 90% CI 2-sided [41.37 to 78.46] — Relative Bioavailability (%) based on CmaxSS for of GSP304 in comparison to SPIRIVA RESPIMAT
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; [analysis description as in outcome 1, analysis 1]; Test type: Other — ANOVA; LS mean ratio (%) = 155.80, 90% CI 2-sided [111.88 to 216.99] — Relative Bioavailability (%) based on CmaxSS for of GSP304 in comparison to SPIRIVA RESPIMAT

2. Primary Outcome: Relative Bioavailability of Tiotropium With GSP 304 in Comparison to SPIRIVA RESPIMAT 5 μg Based on AUC0-tauSS
Description: The PK endpoint in plasma to assess the relative bioavailability was area under the plasma concentration-time curve of tiotropium over the dosing interval at steady state (AUC0-tauSS)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: h*pg/mL
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 26 | 29 | 26 | 26
h*pg/mL | 22.90 (1.130) | 49.10 (1.123) | 122.00 (1.130) | 57.70 (1.130)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; GSP 304 vs SPIRIVA RESPIMAT 5 μg comparison for relative bioavailability data based on AUC0-tauSS was tested and the estimated treatment ratios for the treatment comparisons was presented; Test type: Other — ANOVA; LS mean ratio (%) = 39.70, 90% CI 2-sided [29.79 to 52.87] — Relative Bioavailability (%) based on AUC0-tauSS for of GSP304 in comparison to SPIRIVA RESPIMAT
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; [analysis description as in outcome 2, analysis 1]; Test type: Other — ANOVA; LS mean ratio (%) = 85.20, 90% CI 2-sided [64.43 to 112.64] — Relative Bioavailability (%) based on AUC0-tauSS for of GSP304 in comparison to SPIRIVA RESPIMAT
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; [analysis description as in outcome 2, analysis 1]; Test type: Other — ANOVA; LS mean ratio (%) = 211.50, 90% CI 2-sided [158.80 to 281.80] — Relative Bioavailability (%) based on AUC0-tauSS for of GSP304 in comparison to SPIRIVA RESPIMAT

3. Primary Outcome: Change From Baseline (Day 1) in Trough FEV1 at 24 Hours After the Last Dose of Treatment on Day 21 in Comparison to Placebo.
Description: Change from baseline (Day 1) at Day 21 (Week 3) in trough FEV1 response at approximately 24 hours after the last dose (average of 23 hours 15 minutes and 23 hours 45 minutes postdose measurements), in comparison with placebo.
Time Frame: 21 days (Pre- dose trough FEV1 is mean FEV1 at -45 mins and -15 mins pre-morning dose at Day 1. Trough FEV1 is mean FEV1 obtained 23 hrs 15 mins and 23 hrs 45 mins post-morning dose of day 21).
Measure: Mean (Standard Error); unit: L
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 30 | 32 | 31 | 32 | 30
L | 0.14 (0.04) | 0.10 (0.04) | 0.09 (0.04) | 0.08 (0.04) | 0.14 (0.04)
Statistical Analysis 1: Comparison: GSP304 10 μg vs Placebo; GSP 304 vs Placebo comparison for change from baseline in trough FEV1 was tested at 0.05 significance level; Test type: Superiority; p = 0.228, MMRM; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.04 to 0.17]
Statistical Analysis 2: Comparison: GSP304 20 μg vs Placebo; GSP 304 vs Placebo comparison for change from baseline in trough FEV1 was tested at 0.05 significance level; Test type: Superiority; p = 0.655, MMRM; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.08 to 0.13]
Statistical Analysis 3: Comparison: GSP304 40 μg vs Placebo; GSP 304 vs Placebo comparison for change from baseline in trough FEV1 was tested at 0.05 significance level; Test type: Superiority; p = 0.894, MMRM; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.10 to 0.11]
Statistical Analysis 4: Comparison: Placebo vs SPIRIVA RESPIMAT 5 μg; SPIRIVA RESPIMAT 5 μg vs Placebo comparison for change from baseline in trough FEV1 was tested at 0.05 significance level; Test type: Superiority; p = 0.260, MMRM; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.04 to 0.16]

4. Secondary Outcome: Amount (Aetau) (Cumulative Amount of Unchanged Drug Excreted Into the Urine Over the Dosing Interval) of Tiotropium Excreted in Urine Over the Dosing Interval on Day 1
Description: Descriptive statistics for tiotropium urine PK parameter - Amount (Aetau) of tiotropium excreted in urine over the dosing interval on Day 1
Time Frame: Day 1
Population: Overall Number of Participants Analyzed is the number of subjects with data in the Pharmacokinetic Analysis Set (PKAS). PKAS included all subjects who were randomized, received at least 1 dose of study drug, and had at least 1 quantifiable PK sample and did not have exclusionary major protocol deviations.
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 25 | 23 | 24 | 19
pg | 138600 (76830) | 336100 (233800) | 602900 (422400) | 247400 (219600)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; The mean amount of tiotropium excreted in urine over the dosing interval on Day 1 for GSP304 10 μg was (Geo mean: 108200 pg) and for SPIRIVA RESPIMAT 5 μg was (Geo mean: 120300 pg)
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; The mean amount of tiotropium excreted in urine over the dosing interval on Day 1 for GSP304 20 μg was (Geo mean: 263100 pg) and for SPIRIVA RESPIMAT 5 μg was (Geo mean: 120300 pg)
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; The mean amount of tiotropium excreted in urine over the dosing interval on Day 1 for GSP304 40 μg was (Geo mean: 438300 pg) and for SPIRIVA RESPIMAT 5 μg was (Geo mean: 120300 pg)

5. Secondary Outcome: Amount (Aetau) of Tiotropium Excreted in Urine Over the Dosing Interval on Day 21
Description: Descriptive statistics for tiotropium urine PK parameter - Amount (Aetau) of Tiotropium Excreted in Urine Over the Dosing Interval on Day 21
Time Frame: Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 26 | 29 | 26 | 25
pg | 375400 (286900) | 647100 (460000) | 1611000 (1013000) | 775500 (458000)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; The mean amount of tiotropium excreted in urine over the dosing interval on Day 21 for GSP304 10 μg was (Geo mean: 293700 pg) and for SPIRIVA RESPIMAT 5 μg was (Geo mean: 620200 pg)
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; The mean amount of tiotropium excreted in urine over the dosing interval on Day 21 for GSP304 20 μg was (Geo mean: 436500 pg) and for SPIRIVA RESPIMAT 5 μg was (Geo mean: 620200 pg)
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; The mean amount of tiotropium excreted in urine over the dosing interval on Day 21 for GSP304 40 μg was (Geo mean: 1249000 pg) and for SPIRIVA RESPIMAT 5 μg was (Geo mean: 620200 pg)

6. Secondary Outcome: Fraction of Dose (Fe) of Tiotropium Excreted in Urine Over the Dosing Interval on Day 1
Description: Descriptive statistics for tiotropium urine PK parameter - Fraction of dose (Fe) of tiotropium excreted in urine over the dosing interval on Day 1
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 25 | 23 | 24 | 19
percentage of dose | 1.386 (0.7683) | 1.681 (1.169) | 1.507 (1.056) | 4.948 (4.391)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 10 μg, the geometric mean Fe (%) eliminated in urine was 1.082% on Day 1 and for SPIRIVA RESPIMAT 5 μg, the geometric mean Fe (%) eliminated in urine was 2.407% on Day 1
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 20 μg, the geometric mean Fe (%) eliminated in urine was 1.316% on Day 1 and for SPIRIVA RESPIMAT 5 μg, the geometric mean Fe (%) eliminated in urine was 2.407% on Day 1
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 40 μg, the geometric mean Fe (%) eliminated in urine was 1.096% on Day 1 and for SPIRIVA RESPIMAT 5 μg, the geometric mean Fe (%) eliminated in urine was 2.407% on Day 1

7. Secondary Outcome: Fraction of Dose (Fe) of Tiotropium Excreted in Urine Over the Dosing Interval on Day 21
Description: Descriptive statistics for tiotropium urine PK parameter-Fraction of Dose (Fe) of Tiotropium Excreted in Urine Over the Dosing Interval on Day 21
Time Frame: Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 26 | 29 | 26 | 25
percentage of dose | 3.754 (2.869) | 3.236 (2.300) | 4.026 (2.532) | 15.51 (9.161)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 10 μg, the geometric mean Fe (%) eliminated in urine was 2.937% on Day 21 and for SPIRIVA RESPIMAT 5 μg, the geometric mean Fe (%) eliminated in urine was 12.4% on Day 21
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 20 μg, the geometric mean Fe (%) eliminated in urine was 2.183% on Day 21 and for SPIRIVA RESPIMAT 5 μg, the geometric mean Fe (%) eliminated in urine was 12.4% on Day 21
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 40 μg, the geometric mean Fe (%) eliminated in urine was 3.123% on Day 21 and for SPIRIVA RESPIMAT 5 μg, the geometric mean Fe (%) eliminated in urine was 12.4% on Day 21

8. Secondary Outcome: Peak Concentrations During the Dosing Interval (Cmax) on Day 1
Description: Descriptive statistics for tiotropium plasma PK parameters - (Cmax) on Day 1
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 28 | 27 | 28 | 22
pg/mL | 2.632 (1.690) | 7.119 (7.368) | 14.06 (11.98) | 10.25 (7.944)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 10 μg, geometric mean Cmax of tiotropium was 2.191 pg/mL and for SPIRIVA RESPIMAT 5 μg, geometric mean Cmax of tiotropium was 7.327 pg/mL on Day 1
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 20 μg, geometric mean Cmax of tiotropium was 4.796 pg/mL and for SPIRIVA RESPIMAT 5 μg, geometric mean Cmax of tiotropium was 7.327 pg/mL on Day 1
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 40 μg, geometric mean Cmax of tiotropium was 10.2 pg/mL and for SPIRIVA RESPIMAT 5 μg, geometric mean Cmax of tiotropium was 7.327 pg/mL on Day 1

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUC0-tau) on Day 1
Description: Descriptive statistics for tiotropium plasma PK parameter - Area under the plasma concentration-time curve over the dosing interval (AUC0-tau) on Day 1
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 27 | 26 | 27 | 22
pg*h/mL | 10.65 (7.049) | 22.94 (13.09) | 52.11 (34.7) | 22.64 (10.69)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 10 μg, geometric mean AUC0-tau of tiotropium was 8.597 pg*h/mL and for SPIRIVA RESPIMAT 5 μg, geometric mean AUC0-tau of tiotropium was 19.59 pg*h/mL on Day 1
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 20 μg, geometric mean AUC0-tau of tiotropium was 18.00 pg*h/mL and for SPIRIVA RESPIMAT 5 μg, geometric mean AUC0-tau of tiotropium was 19.59 pg*h/mL on Day 1
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 40 μg, geometric mean AUC0-tau of tiotropium was 42.69 pg*h/mL and for SPIRIVA RESPIMAT 5 μg, geometric mean AUC0-tau of tiotropium was 19.59 pg*h/mL on Day 1

10. Secondary Outcome: Time of Peak Drug Concentration Over the Dosing Interval (Tmax) on Day 1
Description: Descriptive statistics for tiotropium plasma PK parameter - Time of peak drug concentration over the dosing interval (tmax) on Day 1
Time Frame: Day 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 28 | 27 | 28 | 22
hour | 0.067 [0.03 to 0.18] | 0.100 [0.03 to 8.02] | 0.108 [0.03 to 0.75] | 0.100 [0.03 to 3.98]

11. Secondary Outcome: Time of Peak Drug Concentration Over the Dosing Interval (Tmax) on Day 21
Description: Descriptive statistics for tiotropium plasma PK parameter - Time of peak drug concentration over the dosing interval (tmax) on Day 21
Time Frame: Day 21
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 26 | 30 | 26 | 26
hour | 0.075 [0.03 to 0.25] | 0.150 [0.04 to 16.00] | 0.108 [0.05 to 1.00] | 0.100 [0.03 to 0.75]

12. Secondary Outcome: Average Concentration During a Dosing Interval at Steady State (CavSS) on Day 21
Description: Descriptive statistics for tiotropium plasma PK parameter - Average concentration during a dosing interval at steady state (CavSS) on day 21
Time Frame: Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 26 | 30 | 26 | 26
pg/mL | 1.120 (0.8301) | 2.436 (1.623) | 6.273 (4.052) | 2.725 (1.289)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 10 μg, the geometric mean CavSS was 0.9536 pg/mL on Day 21 and for SPIRIVA RESPIMAT 5 μg, the CavSS was 2.403 pg/mL on Day 21
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 20 μg, the geometric mean CavSS was 1.998 pg/mL on Day 21 and for SPIRIVA RESPIMAT 5 μg, the CavSS was 2.403 pg/mL on Day 21
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; For GSP304 40 μg, the geometric mean CavSS was 5.083 pg/mL on Day 21 and for SPIRIVA RESPIMAT 5 μg, the CavSS was 2.403 pg/mL on Day 21

13. Secondary Outcome: Accumulation Ratio Rac(Auc)
Description: Descriptive statistics for tiotropium plasma PK parameter-Accumulation ratio Rac(auc). Rac(auc) was calculated as AUC0-tauSS/AUC0-tau.
Time Frame: Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 26 | 26 | 25 | 25
ratio | 2.966 (1.561) | 5.328 (13.53) | 3.667 (2.873) | 3.699 (2.897)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; Upon repeat dosing, tiotropium had accumulated by Day 21 with a geometric mean accumulation ratio (Rac) based on AUC of 2.617 for GSP304 10 μg and 2.815 for SPIRIVA RESPIMAT 5 μg
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; Upon repeat dosing, tiotropium had accumulated by Day 21 with a geometric mean accumulation ratio (Rac) based on AUC of 2.522 for GSP304 20 μg and 2.815 for SPIRIVA RESPIMAT 5 μg
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; Upon repeat dosing, tiotropium had accumulated by Day 21 with a geometric mean accumulation ratio (Rac) based on AUC of 2.926 for GSP304 40 μg and 2.815 for SPIRIVA RESPIMAT 5 μg

14. Secondary Outcome: Accumulation Ratio Rac(Cmax)
Description: Descriptive statistics for tiotropium plasma PK parameter-Accumulation ratio Rac(cmax). Rac(Cmax) was calculated as CmaxSS/Cmax.
Time Frame: Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 26 | 29 | 26 | 25
ratio | 2.063 (0.7187) | 3.492 (7.436) | 2.622 (2.059) | 2.835 (2.612)
Statistical Analysis 1: Comparison: GSP304 10 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; Upon repeat dosing, tiotropium had accumulated by Day 21 with a geometric mean accumulation ratio (Rac) based on Cmax of 1.944 for GSP304 10 μg and 1.929 for SPIRIVA RESPIMAT 5 μg
Statistical Analysis 2: Comparison: GSP304 20 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; Upon repeat dosing, tiotropium had accumulated by Day 21 with a geometric mean accumulation ratio (Rac) based on Cmax of 1.808 for GSP304 20 μg and 1.929 for SPIRIVA RESPIMAT 5 μg
Statistical Analysis 3: Comparison: GSP304 40 μg vs SPIRIVA RESPIMAT 5 μg; Test type: Other; Upon repeat dosing, tiotropium had accumulated by Day 21 with a geometric mean accumulation ratio (Rac) based on Cmax of 2.125 for GSP304 40 μg and 1.929 for SPIRIVA RESPIMAT 5 μg

15. Secondary Outcome: Change From Baseline in Peak FEV1 Within 12 Hours Post-dose on Day 1
Description: The least square mean change from baseline to peak FEV1 within 12 hours postdose on Day 1. Change from baseline in peak FEV1 within 12 hours postdose on Day 1 was derived from the serial readings taken through 12 hours postdose and calculating the change from baseline.
Time Frame: Day 1 (Pre-dose FEV1 at -45 mins and 15 mins prior to dosing on Day 1. On Day 1 FEV1 at post-dose at 5 mins ±3, 15 mins ±2, 30 mins ±5, 60 mins, 90 mins, and 2 hours; and post-dose at 4, 6, 8, 10, 12 hours after the morning dose).
Population: Full Analysis Set (FAS) included all subjects who were randomized, had received at least 1 dose of study drug and had at least 1 post-baseline PD assessment.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 30 | 32 | 31 | 32 | 30
Litre | 0.34 (0.03) | 0.38 (0.03) | 0.33 (0.04) | 0.21 (0.03) | 0.38 (0.03)
Statistical Analysis 1: Comparison: GSP304 10 μg vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.04 to 0.21]
Statistical Analysis 2: Comparison: GSP304 20 μg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.08 to 0.26]
Statistical Analysis 3: Comparison: GSP304 40 μg vs Placebo; Test type: Superiority; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.03 to 0.21]
Statistical Analysis 4: Comparison: Placebo vs SPIRIVA RESPIMAT 5 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.08 to 0.26]

16. Secondary Outcome: Change From Baseline in Peak FEV1 Within 12 Hours Post-dose on Day 21
Description: The least square mean change from baseline to peak FEV1 within 12 hours postdose on Day 21. Change from baseline in peak FEV1 within 12 hours postdose on Day 21 was derived from the serial readings taken through 12 hours postdose and calculating the change from baseline.
Time Frame: Day 21(Pre-dose FEV1 at -45 mins and 15 mins prior to dosing on Day 21. On Day 21, FEV1 at post-dose at 5 mins ±3, 15 mins ±2, 30 mins ±5, 60 mins, 90 mins, and 2 hours; and post-dose at 4, 6, 8, 10, 12 hours after the morning dose).
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 30 | 32 | 31 | 32 | 30
Litre | 0.37 (0.04) | 0.34 (0.04) | 0.31 (0.04) | 0.20 (0.04) | 0.37 (0.04)
Statistical Analysis 1: Comparison: GSP304 10 μg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.08 to 0.28]
Statistical Analysis 2: Comparison: GSP304 20 μg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.05 to 0.25]
Statistical Analysis 3: Comparison: GSP304 40 μg vs Placebo; Test type: Superiority; p = 0.032, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [0.01 to 0.21]
Statistical Analysis 4: Comparison: Placebo vs SPIRIVA RESPIMAT 5 μg; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.07 to 0.27]

17. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) on Day 1
Description: Least Square Mean change from baseline in forced vital capacity (FVC) to end of Day 1.
Time Frame: Day 1 (Pre-dose FVC at -45 mins and 15 mins prior to dosing on Day 1. Postdose timing were relative to the end of dosing.The window for 1 hour spirometry and thereafter was ±5 minutes).
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 29 | 32 | 31 | 31 | 30
Litre | 0.21 (0.05) | 0.21 (0.05) | 0.18 (0.05) | 0.13 (0.05) | 0.16 (0.05)
Statistical Analysis 1: Comparison: GSP304 10 μg vs Placebo; Test type: Superiority; p = 0.166, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.04 to 0.21]
Statistical Analysis 2: Comparison: GSP304 20 μg vs Placebo; Test type: Superiority; p = 0.182, Mixed Models Analysis; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.04 to 0.21]
Statistical Analysis 3: Comparison: GSP304 40 μg vs Placebo; Test type: Superiority; p = 0.401, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.07 to 0.17]
Statistical Analysis 4: Comparison: Placebo vs SPIRIVA RESPIMAT 5 μg; Test type: Superiority; p = 0.574, Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.09 to 0.16]

18. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) on Day 21
Description: Least Square Mean change from baseline in forced vital capacity (FVC) to end of Day 21
Time Frame: Day 21 (Pre-dose FVC at -45 mins and 15 mins prior to dosing on Day 21. Postdose timing were relative to the end of dosing. The window for 1 hour spirometry and thereafter was ±5 minutes).
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 29 | 32 | 31 | 31 | 30
Litre | 0.16 (0.06) | 0.10 (0.06) | 0.11 (0.06) | 0.11 (0.06) | 0.16 (0.06)
Statistical Analysis 1: Comparison: GSP304 10 μg vs Placebo; Test type: Superiority; p = 0.493, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.10 to 0.21]
Statistical Analysis 2: Comparison: GSP304 20 μg vs Placebo; Test type: Superiority; p = 0.864, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.17 to 0.14]
Statistical Analysis 3: Comparison: GSP304 40 μg vs Placebo; Test type: Superiority; p = 0.978, Mixed Models Analysis; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.16 to 0.15]
Statistical Analysis 4: Comparison: Placebo vs SPIRIVA RESPIMAT 5 μg; Test type: Superiority; p = 0.500, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.10 to 0.20]

19. Secondary Outcome: Change From Baseline in Time-normalized Area Under the Curve for FEV1 Measured Over 12 Hours on Day 1
Description: Least Square Mean (SE) change from baseline in time-normalized area under the curve for FEV1 measured over 12 hours on Day 1.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 29 | 32 | 31 | 31 | 30
Litre | 0.22 (0.03) | 0.24 (0.03) | 0.24 (0.03) | 0.10 (0.03) | 0.26 (0.03)
Statistical Analysis 1: Comparison: GSP304 10 μg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.04 to 0.20]
Statistical Analysis 2: Comparison: GSP304 20 μg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [0.06 to 0.22]
Statistical Analysis 3: Comparison: GSP304 40 μg vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.06 to 0.21]
Statistical Analysis 4: Comparison: Placebo vs SPIRIVA RESPIMAT 5 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [0.08 to 0.23]

20. Secondary Outcome: Change From Baseline in Time-normalized Area Under the Curve for FEV1 Measured Over 12 Hours on Day 21
Description: Least Square Mean (SE) change from baseline in time-normalized area under the curve for FEV1 Measured Over 12 Hours on Day 21.
Time Frame: as for outcome 16
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg
Number analyzed (Participants) | 29 | 32 | 31 | 31 | 30
Litre | 0.23 (0.04) | 0.17 (0.03) | 0.15 (0.04) | 0.08 (0.04) | 0.23 (0.03)
Statistical Analysis 1: Comparison: GSP304 10 μg vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.06 to 0.24]
Statistical Analysis 2: Comparison: GSP304 20 μg vs Placebo; Test type: Superiority; p = 0.061, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.00 to 0.18]
Statistical Analysis 3: Comparison: GSP304 40 μg vs Placebo; Test type: Superiority; p = 0.140, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.02 to 0.16]
Statistical Analysis 4: Comparison: Placebo vs SPIRIVA RESPIMAT 5 μg; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.06 to 0.24]

ADVERSE EVENTS:
Time Frame: The AEs and SAEs were collected from the time of signing the informed consent form until the end of study and the follow-up contact which was approximately 9 weeks i.e., upto 2 weeks of screening, 2 weeks of run-in period, 3 weeks of treatment and follow up of 2 weeks.
Description: GSP304 placebo: One subject not randomized to study treatment inadvertently received placebo and therefore included in SAF in Placebo arm.
Arm/Group | GSP304 10 μg | GSP304 20 μg | GSP304 40 μg | Placebo | SPIRIVA RESPIMAT 5 μg
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32 | 0/31 | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32 | 0/31 | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 6/32 | 5/31 | 4/33 | 6/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSP304 10 μg (N=30) | GSP304 20 μg (N=32) | GSP304 40 μg (N=31) | Placebo (N=33) | SPIRIVA RESPIMAT 5 μg (N=30)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03118765/SAP_000.pdf
  • Study Protocol (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT03118765/Prot_001.pdf